CLINICAL TRIAL: NCT04457362
Title: A Comparative Study Evaluating the Diagnostic Accuracy of Wrist Arthroscopy Using the NanoScope Compared to Conventional Arthroscopic Instrumentation
Brief Title: Wrist Arthroscopy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-00356
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Wrist Arthropathy

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study, Diagnostic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental Cohort (Experimental): Patients with clinically diagnosed wrist pathology undergoing wrist arthroscopy
  Interventions: Diagnostic Test: Diagnostic Arthroscopy using the Arthrex NanoScope; Diagnostic Test: Diagnostic Arthroscopy using standard arthroscopic instruments

INTERVENTIONS:
Diagnostic Test: Diagnostic Arthroscopy using the Arthrex NanoScope — A diagnostic arthroscopy will be performed with the Arthrex NanoScope.
  Structures evaluated:
  * Radial styloid
  * Proximal scaphoid articular cartilage
  * Scaphoid fossa
  * Radioscaphocapitate (RSC) ligament
  * Long radiolunate (LRL) ligament
  * Short radiolunate (SRL) ligament
  * Scapholunate (SL) ligament
  * Proximal lunate articular cartilage
  * Lunate fossa
  * Triangular fibrocartilage complex (TFCC) The attending performing the diagnostic arthroscopy will make an initial diagnostic assessment based on the presence/location/severity of synovitis, articular cartilage integrity, ligament injury and determine the intended treatment.
Diagnostic Test: Diagnostic Arthroscopy using standard arthroscopic instruments — A diagnostic arthroscopy will be performed with the standard arthroscopic instruments.
  Structures evaluated:
  * Radial styloid
  * Proximal scaphoid articular cartilage
  * Scaphoid fossa
  * Radioscaphocapitate (RSC) ligament
  * Long radiolunate (LRL) ligament
  * Short radiolunate (SRL) ligament
  * Scapholunate (SL) ligament
  * Proximal lunate articular cartilage
  * Lunate fossa
  * Triangular fibrocartilage complex (TFCC) The attending performing the diagnostic arthroscopy will make the final diagnostic assessment based on the presence/location/severity of synovitis, articular cartilage integrity, and ligament injury and determine the final treatment.

SUMMARY:
The purpose of this study is to evaluate the diagnostic efficacy of Arthrex NanoScope compared to conventional arthroscopic instruments. Patients with wrist pathology who are indicated for an arthroscopic procedure will be enrolled pre-operatively after a thorough discussion of the study aims, risks, and benefits. At the time of surgery, under standard conditions, using standard wrist arthroscopy portals, a diagnostic arthroscopy will be performed with the Arthrex Nanoscope. The diagnostic arthroscopy will be performed in a stepwise manner for consistency with notation of pathology and intended intervention. The diagnostic arthroscopy will then be performed with the standard arthroscopic equipment, again noting pathology and final intervention. Post-operatively, diagnostic accuracy, incidence of change in intervention, and surgeon rated ease of use and confidence will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Wrist pathology based on clinical examination/imaging studies undergoing wrist arthroscopy for further evaluation/treatment.
3. Willingness to participate in the study

Exclusion Criteria:

* 1. Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Paksima, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [contact information for PI or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication
Access Criteria: Requests should be directed to ali.azad@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Cohort: Patients with clinically diagnosed wrist pathology undergoing wrist arthroscopy
  Diagnostic Arthroscopy using the Arthrex NanoScope: A diagnostic arthroscopy will be performed with the Arthrex NanoScope.
  Structures evaluated:
  * Radial styloid
  * Proximal scaphoid articular cartilage
  * Scaphoid fossa
  * Radioscaphocapitate (RSC) ligament
  * Long radiolunate (LRL) ligament
  * Short radiolunate (SRL) ligament
  * Scapholunate (SL) ligament
  * Proximal lunate articular cartilage
  * Lunate fossa
  * Triangular fibrocartilage complex (TFCC) The attending performing the diagnostic arthroscopy will make an initial diagnostic assessment based on the presence/location/severity of synovitis, articular cartilage integrity, ligament injury and determine the intended treatment.
  Diagnostic Arthroscopy using standard arthroscopic instruments: A diagnostic arthroscopy will be performed with the standard arthroscopic instruments.
  Structures evaluated:
  * Radial styloid
  * Proximal scaphoid articular cartilage
  * Scaphoid fossa
  * Radioscaphocapitate (RSC) ligament
  * Long radiolunate (LRL) ligament
  * Short radiolunate (SRL) ligament
  * Scapholunate (SL) ligament
  * Proximal lunate articular cartilage
  * Lunate fossa
  * Triangular fibrocartilage complex (TFCC) The attending performing the diagnostic arthroscopy will make the final diagnostic assessment based on the presence/location/severity of synovitis, articular cartilage integrity, and ligament injury and determine the final treatment.
Period: Overall Study
Arm/Group | Experimental Cohort
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Surgeon-Rated Radiocarpal Visualization With Arthrex Nanoscope
Description: Radiocarpal visualization rated on a 5-point scale: (1) - bad; (2) - poor; (3) - fair; (4) - good; (5) - excellent.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 4.95 (0.22)

2. Primary Outcome: Surgeon-Rated Radiocarpal Visualization With Conventional Instrument
Description: Radiocarpal visualization rated on a 5-point scale: (1) - bad; (2) - poor; (3) - fair; (4) - good; (5) - excellent.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 4.75 (1.12)

3. Secondary Outcome: Surgeon-rated Ease of Use of Arthrex NanoScope
Description: Ease of use will be rated on a 5-point scale: (1) - very difficult; (2) - difficult; (3) - neutral; (4) - easy; (5) - very easy.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 4.9 (0.31)

4. Secondary Outcome: Surgeon-rated Ease of Use of Conventional Instrument
Description: as for outcome 3
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 4.75 (1.12)

5. Secondary Outcome: Surgeon-rated Confidence in Arthrex NanoScope Diagnosis
Description: Confidence will be rated on a 5-point scale: (1) - not at all confident; (2) - not very confident; (3) - neutral; (4) - fairly confident; (5) - very confident.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 5 (0)

6. Secondary Outcome: Surgeon-rated Confidence in Conventional Instrument Diagnosis
Description: as for outcome 5
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 4.75 (1.12)

7. Primary Outcome: Surgeon-Rated Midcarpal Visualization With Arthrex Nanoscope
Description: Midcarpal visualization rated on a 5-point scale: (1) - bad; (2) - poor; (3) - fair; (4) - good; (5) - excellent.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 5 (0)

8. Primary Outcome: Surgeon-Rated Midcarpal Visualization With Conventional Instrument
Description: Midcarpal visualization rated on a 5-point scale: (1) - bad; (2) - poor; (3) - fair; (4) - good; (5) - excellent.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Cohort
Number analyzed (Participants) | 20
score on a scale | 3.9 (2.02)

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Experimental Cohort
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04457362/Prot_SAP_000.pdf